CLINICAL TRIAL: NCT06998810
Title: Effect of Cerebellar High-Frequency rTMS in Improving Balance Performance in Multiple Sclerosis Patients
Brief Title: Cerebellar High-Frequency rTMS in Balance of Multiple Sclerosis Patients
Acronym: CRESTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R31/2023; FMASUREC (Other: Faculty of Medicine, Ain Shams University)
Record Dates: First submitted 2025-05-06; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis, cerebellar rTMS, balance in Multiple sclerosis,
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded, placebo-controlled prospective study was conducted at Ain Shams University Hospital. Forty MS patients were recruited from specialized MS clinics and physical medicine and Rehabilitation outpatient clinics. All patients signed and informed written consent. Patients were randomly assigned to one of two groups: Treatment Group (n = 20): received real rTMS over the cerebellar vermis, three times per week for 4 weeks. Control Group (n = 20): received sham rTMS using a placebo program. Both groups participated in an intensive exercise training program. An informed written consent was signed from all participants.
Who Masked: Participant
Masking Description: Participants are single-blinded to group assignment. Those in the active group receive real cerebellar rTMS, while the control group receives sham stimulation using an identical coil setup and sound, but without actual magnetic pulses. The treating clinician administering the rTMS is not blinded, but participants are unaware of their assignment to maintain blinding integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Active Comparator - Real rTMS (Active Comparator): Arm Label: Real rTMS
  Type: Active Comparator
  Description:
  Participants in this group receive real repetitive transcranial magnetic stimulation (rTMS) targeting the cerebellum. Stimulation is delivered using a figure-of-eight coil positioned over the vermis of the cerebellum, at a frequency of 10 Hz, work period 5s, number of trains 25, ITI is 25s. The total number of pulses is 1250 pulses per session.
  Interventions: Device: cerebellar rTMS
- Arm 2: Sham Comparator - Sham rTMS (Sham Comparator): Arm Label: Sham rTMS Type: Sham Comparator
  Description:
  Participants in this group receive sham stimulation using the same rTMS device and setup as the active group. The coil is adjusted to mimic the sound and feel of stimulation without delivering an effective magnetic pulse to the brain. Participants are blinded to their assignment to preserve study integrity.
  Interventions: Device: cerebellar rTMS

INTERVENTIONS:
Device: cerebellar rTMS — Non-invasive magnetic stimulation targeting the cerebellum using a figure of eight coil

SUMMARY:
Background: Multiple Sclerosis (MS) is a chronic autoimmune disease affecting the central nervous system (CNS), leading to progressive motor dysfunction and balance deficits. Objective: To investigate the impact of cerebellar rTMS in improving postural control, balance performance and functional ambulation in individuals with MS.

Forty patients were randomly assigned to receive repetitive transcranial magnetic stimulation (rTMS) over the cerebellum to improve motor function and balance in 40 MS patients. Outcome measures, including the Expanded Disability Status Scale (EDSS), static posturography (COP measures), the International Cooperative Ataxia Rating Scale (ICARS), and the 10-Meter Walk Test (10MWT), were assessed before and after intervention.

DETAILED DESCRIPTION:
Background: Multiple Sclerosis (MS) is a chronic autoimmune disease affecting the central nervous system (CNS), leading to progressive motor dysfunction and balance deficits. Although disease-modifying therapies have advanced, there remains an unmet need for effective treatments that target motor and cognitive impairments. Objective: To investigate the impact of cerebellar rTMS in improving postural control, balance performance, and functional ambulation in individuals with MS. Method: This randomized, single-blinded, placebo-controlled clinical trial evaluated the efficacy of repetitive transcranial magnetic stimulation (rTMS) over the cerebellum in improving motor function and balance in 40 MS patients. Outcome measures, including the Expanded Disability Status Scale (EDSS), static posturography (COP measures), the International Cooperative Ataxia Rating Scale (ICARS), and the 10-Meter Walk Test (10MWT), were assessed before and after intervention.

ELIGIBILITY:
Inclusion criteria:

* Patient age ≥18 years.
* Patients with MS, established by clinical, laboratory, MRI criteria and matched Mc Donald's criteria, McDonald et al, 2006.
* Expanded Disability Status Scale (EDSS) scores between 2.5-5
* Only patients in "remitting" phase were included.
* Informed consent.

Exclusion criteria:

* Factors that prevent patient cooperation understanding that impede proper study participation.
* Disabling medical history as severe or recent heart disease and or severe head trauma.
* Cognitive impairment: <24 points by mini-mental scale. (Folstein MF et al., 1975).
* Diabetic patients.
* Patients with any other comorbidity that can affect balance, e.g, other neurological diseases that can affect posterior column function.
* Contraindications for rTMS:

  1. History of epilepsy.
  2. Metal (implants) in skull/scalp/head or fragments from welding or metalwork.
  3. Implanted device (as spinal cord stimulator, cardiac pacemaker, and cochlear implants).
  4. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Static posturography | 3 years
  Static Posturography: Balance assessment using COP measures under eyes-open (COP-O) and eyes-closed (COP-C) conditions.
International Cooperative Ataxia Rating Scale (ICARS) | 3 years
  International Cooperative Ataxia Rating Scale (ICARS): Quantifies ataxia severity.
Expanded Disability Status Scale (EDSS) | 3 years
  Expanded Disability Status Scale (EDSS): Overall disability in MS

SECONDARY OUTCOMES:
10-Meter Walk Test (10MWT) | 3 years
  put marks at 2, 6,&8 meters. measure the time taken from 2 to 8 meters, neglect the rest

CONTACTS AND LOCATIONS:
Locations (1):
- Shereen Ismail Fawaz, Cairo, Other, Egypt